CLINICAL TRIAL: NCT06900218
Title: A Multicenter, Randomized Controlled Phase III Trial of Sintilimab Combined With Capecitabine Versus Capecitabine Alone as Adjuvant Therapy for High-Risk Locoregionally-advanced Nasopharyngeal Carcinoma
Brief Title: PD-1 Antibody Sintilimab Combined With Capecitabine as Adjuvant Therapy for High-Risk Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-FXY-001-FLK
Record Dates: First submitted 2025-03-20; First posted 2025-03-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — sintilimab; spartalizumab; Capecitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sintilimab Combined with Capecitabine (Experimental)
  Interventions: Drug: Sintilimab; Drug: Capecitabine
- Sintilimab (Active Comparator)
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200 mg, administered on Day 1, every 3 weeks for a total of 9 cycles
  Other Names: IBI308; PD-1 antibody
Drug: Capecitabine — Capecitabine 650 mg/m², taken orally twice daily, continuously from Day 1 to Day 21, every 3 weeks, for a maximum of 1 year.
  Arms: Sintilimab Combined with Capecitabine

SUMMARY:
This study will enroll 664 patients who had completed induction chemotherapy combined with the PD-1 antibody sintilimab treatment followed by concurrent cisplatin-based chemoradiotherapy (no concurrent sintiliamb). Patients will be randomly divided into two groups. One group will receive 9 cycles of sintilimab therapy, while the other group will receive an additional year of capecitabine chemotherapy on top of the sintilimab treatment. The primary endpoints will be event-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years.
* ECOG performance status of 0-1.
* Newly diagnosed nasopharyngeal carcinoma confirmed by pathological examination of the primary lesion.
* Staging is classified as T4N1M0 or T1-4N2-3M0 according to the 9th Edition of the American Joint Committee on Cancer/Union for International Cancer Control (AJCC/UICC) staging system.
* Must have received recommended radical radiochemotherapy and sintilimab: 3 cycles of gemcitabine combined with cisplatin and Sintilimab; radical intensity-modulated radiotherapy with a total dose of 6,996 cGy over 33 fractions, concurrently receiving 2 cycles of cisplatin at 100 mg/m².
* Completed the last radiation treatment within 2 weeks before randomization.
* neutrophil count ≥ 1.5 × 10⁹/L, hemoglobin concentration ≥ 90g/L, platelet count ≥ 100 × 10⁹/L.
* Total bilirubin ≤ 1.5 times the upper limit of normal; AST and/or ALT ≤ 2.5 times the upper limit of normal; creatinine clearance ≥ 50 mL/min.
* Participants must sign an informed consent form and be willing and able to comply with the study's visit, treatment regimen, laboratory tests, and other requirements.
* Female participants of childbearing potential and male participants with fertile partners must agree to use reliable contraception (such as condoms, or physician-recommended contraceptive pills) from screening to one year post-treatment.

Exclusion Criteria:

* Active, known, or suspected autoimmune diseases. Participants with Type I diabetes, hypothyroidism requiring only hormone replacement therapy, or skin diseases (e.g., vitiligo, psoriasis, or alopecia) that do not require systemic treatment can be included.
* Severe immune-related adverse events that occurred during the initial Sintilimab induction treatment, as judged by the investigator, preventing continued adjuvant treatment with Sintilimab.
* Received any non-diagnostic surgeries or other targeted, immune, or biological therapies for nasopharyngeal carcinoma except the recommended radiochemotherapy and Sintilimab treatment before randomization.
* factors affecting oral medication (e.g., swallowing difficulties, chronic diarrhea, bowel obstruction).
* Disease progression post-radical radiotherapy.
* Positive HBsAg with HBV DNA > 200 IU/ml or 1000 copies/ml.
* Positive HCV antibody.
* Received systemic corticosteroids or other immunosuppressive therapy at equivalent doses > 10 mg of prednisone/day within 28 days before informed consent. Patients on systemic corticosteroids ≤ 10 mg of prednisone/day or inhaled/topical corticosteroids can be included. Using corticosteroids to manage or prevent treatment-related toxicity is permissible for inclusion.
* Active tuberculosis. Patients with active tuberculosis within the past year are excluded, even if treated; patients with a history of active tuberculosis over one year ago are also excluded unless they can prove they have undergone standard anti-tuberculosis therapy.
* History of interstitial lung disease.
* Received a live vaccine within 30 days before informed consent or is scheduled to receive one.
* HIV infection.
* Current or previous malignancies, except for adequately treated non-melanoma skin cancer, cervical carcinoma in situ, or papillary thyroid carcinoma.
* Pregnant or breastfeeding women; pregnancy tests should be considered for sexually active women of childbearing potential.
* Other diseases or conditions assessed by the investigator that may jeopardize patient safety or compliance, such as unstable cardiac diseases, renal diseases, chronic hepatitis, poorly controlled diabetes, psychiatric disorders, severely abnormal laboratory results, or other family or social high-risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2033-05-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 3-years
Overall survival (OS) | 5-years

SECONDARY OUTCOMES:
Distant metastasis-free survival (DMFS) | 3-years
Locoregional recurrence-free survival (LRFS) | 3-years
Adverse events (AEs) and serious adverse events (SAEs) | 5-years
Quality of life (QoL) | 5-years
  The change of QoL from randomization to 9 weeks (at the 3rd cycle of adjuvant sintilimab treatment), 1 year, 2 years, 3 years, 4 years, and 5 years after randomization. The EORTC QoL questionnaire-C30 (EORTC QLQ-C30) version 3.0 will be used. This questionnaire comprises 30 questions, 24 aggregated into nine multi-question scales: five functioning scales (e.g., physical), three symptom scales (e.g., fatigue), and one global health status scale. The remaining six single-question (e.g., dyspnoea) scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual of EORTC QLQ-C30.
Event-free survival (EFS) within different subgroups | 3-years
  analyses for EFS will be performed within the following subgroups: Epstein-Barr virus (EBV) DNA (=0 vs. >0copies/ml after radiotherapy), different PD-L1 CPS (0 vs. ≥1), tertiary lymphoid structure (+ vs. -), age, sex, performance status, T category, N category, and stage (II vs. III).
Overall survival (OS) within different subgroups | 5-years
  analyses for OS will be performed within the following subgroups: Epstein-Barr virus (EBV) DNA (=0 vs. >0copies/ml after radiotherapy), different PD-L1 CPS (0 vs. ≥1), tertiary lymphoid structure (+ vs. -), age, sex, performance status, T category, N category, and stage (II vs. III).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China, China

IPD SHARING:
Plan to Share IPD: Yes
Complete de-identified patient data set
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: For 2 years, it started 24 months after the primary trial report was published.
Access Criteria: Authoritative researchers who provide a methodologically sound proposal for individual participant data meta-analysis.